CLINICAL TRIAL: NCT04352556
Title: SARS-CoV-2 Infection in Patients With Hematological Malignancies: the Italian Hematology Alliance
Brief Title: COVID19-hematological Malignancies: the Italian Hematology Alliance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Francesco Passamonti, Principal Investigator, Ospedale di Circolo - Fondazione Macchi
Other Study IDs: HM-COVID19-Italy
Record Dates: First submitted 2020-04-09; First posted 2020-04-20 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2 Infection; Hematological Malignancies
Keywords: Hematological Malignancies; Covid-19; SARS-CoV-2; Italian Hematology Alliance; Leukemia; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective/prospective, cohort, non-interventional observational study. This means that all patients with documented COVID and HM diagnosed between February 2020 and study initiation will compose the retrospective part, while those diagnosed after study approval will enter prospective part.

The total duration of the study will be 12 months.

The study population will must be older than 18 years of age with HM and SARS-CoV-2 infection. All patients with documented SARS-CoV-2 infection (COVID) and history or active hematological malignancies, who refer to any Hematological Unit will be included.

DETAILED DESCRIPTION:
This is a retrospective/prospective, cohort, non-interventional observational study. An informed consensus for the participation is available. In this section we provide informations on sample size and statistical analysis.

In Italy, the projected estimate of complete HM prevalence at Jan 1, 2020 has been established as 48,254 cases for Hodgkin lymphoma, 110.715 cases for non Hodgkin Lymphomas, 67,301 for leukemias, and 25,066 for multiple myeloma (Guzzinati et al, BMC Cancer 2018). The Italian Dipartimento della Protezione Civile website reported (March 23, 2020) that 63,927 cases are currently infected with SARS-CoV-2. No formal sample size calculation was made for this project but, on the basis of data available to date, considering the prevalence of hematological patients in Italy (0.4%) and assuming that these patients have the same risk of contracting COVID-19 as the general population, we supposed to enroll at least 250 patients (at March 24, 2020).

Statistical analyses All data collected will be summarized using appropriate descriptive statistics: absolute and relative frequencies for discrete variables; mean, standard deviation, median and interquartile range for continuous ones. To identify factors significantly associated with composite endpoint, log-binomial regression will be used for modelling risk ratio together with 95% confidence interval estimated.

The least absolute shrinkage and selection operator (LASSO) method will be applied for selecting the factors able to independently predict primary end-point. LASSO selects variables correlates to the measured outcome by shrinking coefficients weights, down to zero for the ones not correlated to outcome. In addition, machine learning techniques will be used for validating results from LASSO. A weight will be assigned to each coefficient of the selected predictors and weights will be summed to produce a total aggregate score. Predictive performance will be assessed through discrimination and calibration. Discrimination indicates how well the model can distinguish individuals with the outcome from those without the outcome. Two, the net reclassification improvement (NRI) will be calculated for assessing the 'net' number of individuals correctly reclassified using "the new model" over a comparator index [i.e., CCI (Charlson Comorbidity Score) or MCS (Multisource Comorbidity Score), or HM-disease specific]. Calibration ascertains the concordance between the model's predictions and observed outcomes, which we evaluated using a calibration plot. Cartographic and geostatistical methods will be used to exploring the spatial patterns of disease. An Exploratory Spatial Data Analysis (ESDA) and the Kriging method will be also applied to describe and model spatial (geographical) pattern.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years of age.
* History of hematological malignancies (acute leukemias, myelodysplastic syndromes, myeloproliferative neoplasms, lymphomas, myeloma).
* Active hematological malignancies (acute leukemias, myelodysplastic syndromes, myeloproliferative neoplasms, lymphomas, myeloma) at any stage/status.
* SARS-CoV-2 positive test (nasopharyngeal, BAL, fecal), documented by Real-Time Reverse Transcriptase (RT)-PCR Diagnostic Panels.

Exclusion Criteria:

* Hematological diseases, other than hematological malignancies.
* SARS-CoV-2 negative test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will must be older than 18 years of age with Hematological malignancies and SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate mortality. | At 2 months from study initiation
  The percentage of HM patients with COVID-19 who died.
To evaluate potential predictive biochemical parameters of mortality. | At 2 months from study initiation
  We will assess the correlation between some biochemical parameters at diagnosis of COVID (i.e. hemoglobin, platelets, lymphocytes, clotting tests, CRP), each on the basis of its specific unit of measure, and mortality.
To evaluate potential predictive HM-related parameters of mortality. | At 2 months from study initiation
  We will assess the correlation between HM-related parameters at diagnosis of COVID [i.e. disease type (leukemia, lymphomas, myeloma), disease status (remission / stable / progression), therapy status (on / off therapy)] and mortality.
To evaluate COVID severity as predictive parameter of mortality. | At 2 months from study initiation
  We will assess the correlation between COVID severity [mild (non-pneumonia and mild pneumonia), severe (dyspnea, respiratory frequency ≥ 30/min, SpO2 ≤ 93%, PaO2/FiO2 < 300 and/or lung infiltrates > 50%) and critical (respiratory failure, septic shock, and/or multiple organ disfunction or failure)] and mortality

SECONDARY OUTCOMES:
Epidemiology of patients with HM infected by SARS-CoV-2with any spectrum of illness severity | At 6 months from study initiation
  Description of the different types of hematological malignancies (WHO criteria) in patients with SARS-CoV-2 infection. All aggregated data will be stratified on the basis of COVID severity: mild (non-pneumonia and mild pneumonia), severe (dyspnea, respiratory frequency ≥ 30/min, SpO2 ≤ 93%, PaO2/FiO2 < 300 and/or lung infiltrates > 50%) and critical disease (respiratory failure, septic shock, and/or multiple organ disfunction or failure)
Definition of complete clinical picture of COVID-19 in HM | At 2 months from study initiation
  Characterization of clinical and biochemical profile of patients with SARS-CoV-2 positivity.
Evolution of HM | At 2 months from study initiation
  Assessment of HM status post SARS-CoV-2 infection stratified as no implication, loss of response, progression of the hematological disease.
To evaluate admission to ICU requiring mechanical ventilation or death per characteristics | At 2 months from study initiation
  Percentage of HM patients being admitted to ICU requiring mechanical ventilation, or death stratified per disease type, status, per off-therapy/on-therapy, per type of therapy (chemo, immunotherapy, cell therapy, stem cell transplant).
Viral dynamics in infected HM patients | At 12 months from study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Passamonti, MD, Principal Investigator — Ospedale di Circolo e Fondazione Macchi, ASST Sette Laghi, Varese, Italy
Locations (78):
- Italy (78):
  - SC Ematologia Ospedale SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - UOC Ematologia, Ospedali Riuniti, Ancona
  - UOC Ematologia e Terapia Cellulare, Ospedale Mazzoni, Ascoli Piceno
  - SC Oncologia Medica, CRO, Aviano
  - SC Ematologia, Policlinico Bari, Bari
  - UOC Ematologia, I.R.C.C.S Istituto Tumori Giovanni Paolo II, Bari
  - SSD Ematologia, Ospedale degli Infermi, Biella
  - UOC Ematologia, Azienda Ospedaliero-Universitaria Policlinico S.Orsola-Malpighi,, Bologna
  - Ematologia e Centro Trapianto Midollo Osseo, Ospedale di Bolzano, Bolzano
  - UO Ematologia e CTMO, ASST Spedali Civili, Brescia
  - UOC Onco-Ematologia ASST Valle Olona, Busto Arsizio
  - SC Ematologia e CTMO AZIENDA OSPEDALIERA "G. BROTZU" - OSPEDALE ONCOLOGICO BUSINCO, Cagliari
  - UOC Ematologia, AOU Policlinico Vittorio Emanuele, Catania
  - Ematologia, Ospedale Valduce, Como
  - UOC Ematologia, Azienda Ospedaliera di Cosenza, Cosenza
  - UO Ematologia e CTMO, ASST Cremona, Cremona
  - SC Ematologia Ospedale S. Croce, Cuneo
  - UOC, Ematologia Azienda Ospedaliero Universitaria Arcispedale S. Anna, Ferrara
  - S.O.D. Ematologia, Azienda Ospedaliero Universitaria Careggi, Florence
  - UOC Ematologia, Policlinico Ospedali Riuniti, Foggia
  - IRST-IRCC di Meldola, Forlì
  - UO Ematologia, Ospedale Policlinico S.Martino IRCCS, Genova
  - UO Ematologia, Ospedale Policlinico San Martino, Genova
  - UOC di Ematologia e Trapianto di Cellule Staminali, P.O. Vito Fazzi, Lecce
  - UOC di Ematologia, Ospedale di Legnano, Legnano
  - UO Dipartimento di Ematologia, USL 6, Livorno
  - UOC Oncologia ASST Lodi, Lodi
  - UOC Ematologia Azienda Ospedaliera Universitaria "G.Martino", Messina
  - UO Ematologia, Ospedale dell'Angelo di Mestre, Mestre
  - Ematologia, IEO, Milan
  - SC Ematologia, Istituto Nazionale dei Tumori, Milan
  - SC Ematologia, Ospedale Niguarda, Milan
  - UO Ematologia, IRCCS Ospedale San Raffaele, Milan
  - UO Servizio di Ematologia e Medicina Trasfusionale, Ospedale Luigi Sacco, Milan
  - UOC Ematologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - UO Ematologia Policlinico di Modena, Modena
  - UOC Ematologia, Ospedale S. Gerardo, Monza
  - SC Ematologia Istituto Nazionale Tumori - IRCCS "Fondazione G. Pascale",, Napoli
  - UOC Ematologia e Trapianti di Midollo, AOU Federico II, Napoli
  - UOC Ematologia, Ospedale Antonio Cardarelli, Napoli
  - UOC Ematologia, Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - Ospedale san Luigi Gonzaga, Orbassano
  - Ematologia Azienda Ospedaliera di Padova, Padua
  - UO Ematologia, Policlinico Paolo Giaccone, Palermo
  - UOC Ematologia e CTMO, Azienda Ospedaliero-Universitaria di Parma, Parma
  - SC Ematologia, Fondazione IRCCS Policlinico San Matteo, Pavia
  - SC Ematologia e Trapianto di Midollo Osseo, Azienda Ospedaliera di Perugia, Perugia
  - UO Ematologia e CTMO, Azienda Ospedaliera Ospedali Riuniti, Pesaro
  - UOC di Ematologia, Ospedale Civile Spirito Santo, Pescara
  - UO Ematologia e CTMO, Presidio Ospedaliero di Piacenza, Piacenza
  - UO Ematologia, AOU Pisana- Santa Chiara, Pisa
  - UO Ematologia dell'Ospedale Santa Maria delle Croci, Ravenna
  - UOC Ematologia, Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - SC Ematologia, Arcispedale Santa Maria Nuova, Reggio Emilia
  - UO Ematologia, Ospedale Infermi, Rimini
  - AOU Azienda Ospedaliera Universitaria Sant'Andrea, Roma
  - IFO - Ematologia e Trapianto Cellule -Istituto Nazionale del Cancro di Regina Elena, Roma
  - SC Ematologia, Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - UO Ematologia e Trapianti di Cellule Staminali, A.O. S. Camillo-Forlanini, Roma
  - UO Ematologia, Policlinico Tor Vergata, Roma
  - UOC Ematologia e trapianto di cellule staminali, Policlinico Universitario Campus Bio-Medico, Roma
  - UOC Ematologia Policlinico Umberto I, Roma
  - UOC Ematologia, Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - UOC Ematologia- Azienda Ospedaliera San Giovanni Addolorata, Roma
  - UO Ematologia, Istituto Clinico Humanitas, Rozzano
  - UOC Ematologia e centro trapianti cellule staminali emopoietiche, AOU San Giovanni Di Dio e Ruggi D'aragona, Salerno
  - Ematologia ASL Imperiese, Sanremo
  - Medicina Interna ed Ematologia, Asl 1, Savona
  - UOC Ematologia, Policlinico Santa Maria alle Scotte, Siena
  - UOC Ematologia e Trapianto Midollo Osseo, Ospedale S. G. Moscati, Taranto
  - SCDU Ematologia e terapie cellulari, Ospedale Mauriziano Umberto I, Torino
  - UO Ematologia, Ospedale Universitario Molinette San Giovanni Battista, Torino
  - UO Ematologia, Ospedale Civili Ca' Foncello, Treviso
  - SC Ematologia, Azienda sanitaria universitaria Giuliano Isontina, Trieste
  - Clinica Ematologia, Azienda Ospedaliera-Universitaria Santa Maria della Misericordia, Udine
  - UOC Ematologia, ASST Sette Laghi, Osp. Di Circolo e Fondazione Macchi, Varese
  - UOC Ematologia, Azienda Ospedaliera Integrata di Verona, Verona
  - UOC Ematologia, Ospedale San Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] Xia Y, Jin R, Zhao J, Li W, Shen H. Risk of COVID-19 for patients with cancer. Lancet Oncol. 2020 Apr;21(4):e180. doi: 10.1016/S1470-2045(20)30150-9. Epub 2020 Mar 3. No abstract available. PMID 32142622
- [Background] Wang H, Zhang L. Risk of COVID-19 for patients with cancer. Lancet Oncol. 2020 Apr;21(4):e181. doi: 10.1016/S1470-2045(20)30149-2. Epub 2020 Mar 3. No abstract available. PMID 32142621
- [Background] Corrao G, Rea F, Di Martino M, De Palma R, Scondotto S, Fusco D, Lallo A, Belotti LMB, Ferrante M, Pollina Addario S, Merlino L, Mancia G, Carle F. Developing and validating a novel multisource comorbidity score from administrative data: a large population-based cohort study from Italy. BMJ Open. 2017 Dec 26;7(12):e019503. doi: 10.1136/bmjopen-2017-019503. PMID 29282274
- [Derived] Visco C, Marcheselli L, Mina R, Sassone M, Guidetti A, Penna D, Cattaneo C, Bonuomo V, Busca A, Ferreri AJM, Bruna R, Petrucci L, Cairoli R, Salvini M, Bertu L, Ladetto M, Pilerci S, Pinto A, Ramadan S, Marchesi F, Cavo M, Arcaini L, Coviello E, Romano A, Musto P, Massaia M, Fracchiolla N, Marchetti M, Scattolin A, Tisi MC, Cuneo A, Della Porta M, Trentin L, Turrini M, Gherlinzoni F, Tafuri A, Galimberti S, Bocchia M, Cardinali V, Cilloni D, Corso A, Armiento D, Rigacci L, La Barbera EO, Gambacorti-Passerini C, Visani G, Vallisa D, Venditti A, Selleri C, Conconi A, Tosi P, Lanza F, Candoni A, Krampera M, Corradini P, Passamonti F, Merli F; ITA-HEMA-COV investigators. A prognostic model for patients with lymphoma and COVID-19: a multicentre cohort study. Blood Adv. 2022 Jan 11;6(1):327-338. doi: 10.1182/bloodadvances.2021005691. PMID 34644385
- [Derived] Passamonti F, Cattaneo C, Arcaini L, Bruna R, Cavo M, Merli F, Angelucci E, Krampera M, Cairoli R, Della Porta MG, Fracchiolla N, Ladetto M, Gambacorti Passerini C, Salvini M, Marchetti M, Lemoli R, Molteni A, Busca A, Cuneo A, Romano A, Giuliani N, Galimberti S, Corso A, Morotti A, Falini B, Billio A, Gherlinzoni F, Visani G, Tisi MC, Tafuri A, Tosi P, Lanza F, Massaia M, Turrini M, Ferrara F, Gurrieri C, Vallisa D, Martelli M, Derenzini E, Guarini A, Conconi A, Cuccaro A, Cudillo L, Russo D, Ciambelli F, Scattolin AM, Luppi M, Selleri C, Ortu La Barbera E, Ferrandina C, Di Renzo N, Olivieri A, Bocchia M, Gentile M, Marchesi F, Musto P, Federici AB, Candoni A, Venditti A, Fava C, Pinto A, Galieni P, Rigacci L, Armiento D, Pane F, Oberti M, Zappasodi P, Visco C, Franchi M, Grossi PA, Bertu L, Corrao G, Pagano L, Corradini P; ITA-HEMA-COV Investigators. Clinical characteristics and risk factors associated with COVID-19 severity in patients with haematological malignancies in Italy: a retrospective, multicentre, cohort study. Lancet Haematol. 2020 Oct;7(10):e737-e745. doi: 10.1016/S2352-3026(20)30251-9. Epub 2020 Aug 13. PMID 32798473